CLINICAL TRIAL: NCT03847337
Title: Can Novel Telemedicine Tools Reduce Disparities Related to Early Identification of Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Zachary Warren, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 190152; 1R21MH118539-01 (NIH)
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Results first posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-10

CONDITIONS: Autism Spectrum Disorder; Developmental Delay
Keywords: telemedicine
MeSH Terms: conditions — Autism Spectrum Disorder; Learning Disabilities

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New to diagnosis (Experimental): We will test two telemedicine tools with children who have not been previously diagnosed with autism or developmental delay. The two telemedicine tools are the Screening Tool for Autism in Toddlers (TELE-STAT) and the Autism Spectrum Disorder (ASD-PEDS).
  Interventions: Other: Telehealth-Screening Tool for Autism in Toddlers (STAT); Other: Telehealth-Autism Spectrum Disorder-Pediatrics (ASD-PEDS)
- Previously diagnosed (Experimental): We will test two telemedicine tools with children who have been previously diagnosed with autism or developmental delay. The two telemedicine tools are the Screening Tool for Autism in Toddlers (TELE-STAT) and the Autism Spectrum Disorder (ASD-PEDS).
  Interventions: Other: Telehealth-Screening Tool for Autism in Toddlers (STAT); Other: Telehealth-Autism Spectrum Disorder-Pediatrics (ASD-PEDS)

INTERVENTIONS:
Other: Telehealth-Screening Tool for Autism in Toddlers (STAT) — Structured autism screening tool
Other: Telehealth-Autism Spectrum Disorder-Pediatrics (ASD-PEDS) — Semi-structured autism screening tool

SUMMARY:
In this study, the investigators are trying to find new ways to screen for autism spectrum disorder (ASD) in young children. The investigators want to see if people like pediatricians can screen children for ASD while a psychologist watches on a monitor. The investigators are testing two screening tools. The investigators want to see if they are good at identifying children with ASD and children without ASD. The investigators hope this research will make it easier for families to get answers when there are concerns for ASD.

DETAILED DESCRIPTION:
The investigators will evaluate and compare two telemedicine assessment tools (TELE-STAT and TELE-ASD-PEDS) that could allow parents or naive providers in remote locations to complete an Autism Spectrum Disorder (ASD) risk assessment via telemedicine consultation via an expert psychologist. These tools will be low cost, compliant with privacy rules, easily deployed in community practice settings, and explicitly designed to work within paradigms that may be pragmatically and financially viable for systems of care housing remote clinicians. These telemedicine tools could provide methodologies wherein children could be rapidly linked to and appropriately assessed by ASD experts within practice locations where the children are currently receiving care. In turn, these children, who without such assessment may wait months or over a year in many circumstances to access assessments and interventions, may be able to receive appropriate ASD assessments within days or weeks of screening/surveillance concerns within practice settings where the children are already accessing and familiar with (i.e., minimizing loss to referral and follow-up)

ELIGIBILITY:
Inclusion Criteria:

* Children who have been diagnosed with autism or developmental delay

Exclusion Criteria:

* Children with genetic disorders
* Children with medical complexities, such as blindness or deafness
* Children whose families do not speak English

Ages: 15 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary E Warren, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ASD-PEDS: We will test the ASD-PEDS with children who have not been previously diagnosed with autism or developmental delay.
  Telehealth-Autism Spectrum Disorder-Pediatrics (ASD-PEDS): Semi-structured autism screening tool
- TELE-STAT: We will test the TELE-STAT with children who have not been previously diagnosed with autism or developmental delay.
  Telehealth-Screening Tool for Autism in Toddlers (STAT): Structured autism screening tool
Period: Overall Study
Arm/Group | ASD-PEDS | TELE-STAT
Started | 73 | 71
Completed | 73 | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASD-PEDS | TELE-STAT | Total
Number analyzed (Participants) | 73 | 71 | 144
Age, Continuous [Median (Full Range); unit: years] | 2.57 [1.71 to 3.02] | 2.58 [1.39 to 2.99] | 2.57 [1.39 to 3.02]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 15 | 41
  Male | 47 | 56 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 56 | 63 | 119
  Unknown or Not Reported | 10 | 5 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 11 | 18
  White | 59 | 49 | 108
  More than one race | 3 | 9 | 12
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 73 | 71 | 144

OUTCOME MEASURES:

1. Primary Outcome: Accurate Diagnosis of Autism Via Telemedicine
Description: Number of children who are accurately diagnosed with autism via diagnostic evaluation
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | ASD-PEDS | TELE-STAT
Number analyzed (Participants) | 73 | 71
Participants | 61 | 63

2. Primary Outcome: Accurate Diagnosis of Developmental Delay Via Telemedicine
Description: Number of children who are accurately diagnosed via diagnostic evaluation
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | ASD-PEDS | TELE-STAT
Number analyzed (Participants) | 73 | 71
Participants | 7 | 2

ADVERSE EVENTS:
Time Frame: Day of assessment
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | ASD-PEDS | TELE-STAT
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/71
Other Adverse Events (participants affected / at risk) | 0/73 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT03847337/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT03847337/ICF_001.pdf